CLINICAL TRIAL: NCT06242587
Title: Comparison of Coccygeal Block and Impar Block for the Treatment of Coccydynia
Brief Title: Impar VS Coccygeal Block in the Treatment of Coccidine
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Damla Yürük, medical doctor, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: impar
Record Dates: First submitted 2024-01-13; First posted 2024-02-05 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Coccyx Injury; Coccygeal Body Tumor
Keywords: Coccigodynia; Coccigeal pain treatment; Pericoccigeal nerve block; Impar ganglion block

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Pericoccygeal block (Active Comparator): Patients undergoing pericoccygeal block
  Interventions: Device: Pericoccygeal nerve block
- Group Impar ganglion block (Active Comparator): Patients undergoing impar ganglion block
  Interventions: Procedure: Impar ganglion block

INTERVENTIONS:
Device: Pericoccygeal nerve block — The coccygeal corneas are visualised with a linear probe under ultrasound guidance. The pericoccygeal nerves are located medial to the cornu and a combination of local anaesthetic and dexamethasone is injected.
  Arms: Group Pericoccygeal block
Procedure: Impar ganglion block — The sacrum is visualised with fluoroscopy. A needle is inserted through the sacrococcygeal junction. The optimal image is obtained by administering contrast material. A combination of local anaesthetic and dexamethasone is injected.
  Arms: Group Impar ganglion block

SUMMARY:
The aim of this study was to evaluate the efficacy of coccygeal nerve blockade. Impar sympathetic ganglion blockade is a common treatment method used in coccygeal pain. However, experience with the coccygeal nerve is scarce in the literature. The investigator planned to follow up coccidynia patients who underwent impar sympathetic ganglion blockade and coccygeal nerve blockade for 3 months after the procedure. The investigator's aim is to compare the efficacy of coccygeal nerve blockade with impar blockade.

DETAILED DESCRIPTION:
Patients with coccygeal pain will be evaluated. Patients with organic pathology such as malignancy and infection on imaging and investigations will be excluded. Seventy-four patients diagnosed with traumatic or idiopathic coccidynia will be included in the study. Patients will be randomised by computer programme. Half of them will undergo ultrasound-guided pericoccygeal nerve blockade and the other half will undergo fluoroscopy-guided impar sympathetic ganglion blockade. Pericoccygeal nerve block is performed with the patients lying in the prone position. The sacral horns are visualised using a linear probe. The coccygeal nerves are captured medial to the sacral cornuas and a combination of local anaesthetic and dexamethasone is injected. Impar sympathetic ganglion blockade It is performed in the operating theatre with the patient in the prone position. The sacrum and coccyx are visualised with a lateral view. A needle is inserted through the sacrococcygeal junction and a combination of local anaesthetic and dexamethasone is injected when an optimal image is obtained with contrast material injection. Patients will be evaluated before, 1 and 3 months after the procedure by filling out the Visual analogue scale and PARIS functional coxidynia questionnaire. The investigator who evaluates the patients and collects the data after the procedure will be blinded.

ELIGIBILITY:
Inclusion Criteria:

* Coccygeal pain

Exclusion Criteria:

* Malignite
* Infection
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2024-04-18 (Estimated); Study Completion 2024-05-19 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale | Before treatment, week 4 and week 12
  A Visual Analogue Scale (VAS) is the pain rating scales. Numbers 0-10 represent the severity of the patients' pain. No pain : 0, Most severe pain : 10

SECONDARY OUTCOMES:
PARIS coccidini scale | Before treatment, week 4 and week 12
  Aims to measure functionality. There are options asking whether there is pain during movements such as sitting, standing, walking. the highest value is 10, the lowest value is 0

CONTACTS AND LOCATIONS:
Locations (1):
- Gevher Rabia Genç Perdecioğlu, Ankara, Çankaya, Turkey (Türkiye)